CLINICAL TRIAL: NCT06223074
Title: Towards the Improvement of the Treatment of Acute Relapses in Multiple Sclerosis: A Randomized Double-blind, Non-inferiority Controlled Trial Comparing Intranasal Versus Intravenous Methylprednisolone
Brief Title: Improving the Treatment of Acute Relapses in Multiple Sclerosis Through Intranasal Methylprednisolone Administration
Acronym: IN-DXM-EMRR
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: Instituto Nacional de Neurología y Neurocirugía (Unknown)
Responsible Party: Principal Investigator, Edda Sciutto Conde, Principal Investigator, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BD2012-34CEC
Record Dates: First submitted 2023-04-25; First posted 2024-01-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis Relapsing Remitting; Treatment
Keywords: methylprednisolone; intranasal administration; Multiple Sclerosis Relapsing Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: A prospective, comparative, randomized, controlled study in adult patients with confirmed Relapsing-Remitting Multiple Sclerosis that assits to the hospital with an acute relapse.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Intravenous Methylprednisolone treatment in relapsing-remittent multiple sclerosis (Active Comparator): Intravenous methylprednisolone is the standard treatment for a multiple sclerosis relapse. Thus, 40 randomly enrolled patients aged 18-65 years with relapsing-remitting multiple sclerosis that assist to the hospital and confirmed with a relapse, will be treated with intravenous methylprednisolone, 1000 mg, once a day for 3 days for moderate relapses or 5 days for severe ones.
  A written informed consent will be obtained from each participant or a legal representative whenever the participant could not provide consent.
  Interventions: Other: IV Methylprednisolone administration
- Intranasal Methylprednisolone administration in relapsing-remittent multiple sclerosis (Experimental): Nasal Methylprednisolone Administration For this group, 40 randomly enrolled patients aged 18-65 years with relapsing-remitting multiple sclerosis that assist to the hospital and confirmed with a relapse, will be treated with intranasal methylprednisolone administration (1000 mg once a day for 3 days for moderate relapses or 5 days for severe ones) using a Mucosal Atomization Device (MAD Nasal).
  A written informed consent will be obtained from each participant or a legal representative whenever the participant could not provide consent
  Interventions: Drug: Nasal Methylprednisolone (MT)

INTERVENTIONS:
Other: IV Methylprednisolone administration — Group 1 will receive 1g methylprednisolone IV for 3 or 5 days, according to the severity of the relapse
  Other Names: ST
  Arms: Standard Intravenous Methylprednisolone treatment in relapsing-remittent multiple sclerosis
Drug: Nasal Methylprednisolone (MT) — Group 2 will receive the dose intranasal equivalent to 1g of methylprednisolone for 3 or 5 days according to the severity of the relapse
  Other Names: Nasal MT
  Arms: Intranasal Methylprednisolone administration in relapsing-remittent multiple sclerosis

SUMMARY:
This Clinical Trial evaluates the nasal administration of Methylprednisolone as a treatment strategy for Acute Relapses in Multiple Sclerosis

DETAILED DESCRIPTION:
This is a prospective, comparative, randomized, double-blind study adhered to the principles established by the Helsinki Declaration, including informed consent. Patients with a diagnosis of Relapsing-Remitting Multiple Sclerosis (RRMS) from the National Institute of Neurology and Neurosurgery (INNN) that are coursing with acute recurrency will be included. The recruited patients will be organized into two paired groups of 40 patients each, of which group 1 will receive 1g IV methylprednisolone, and group 2 will receive the intranasal dose equivalent to 1g of IV methylprednisolone. Clinical symptoms will be measured with the Expanded Disability Status Scale (EDSS) and data will be complemented with results of clinical tests, general laboratories and serum concentration of MP and inflammatory markers. Adverse effects in each group will also be identified and quantified. Statistical analysis: descriptive, assumption of normality, bivariate comparison of means and multivariate, in addition to intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Diagnosis of RRMS with an evolution from diagnosis of 3 months to 10 years.
* Kurtzke Expanded Disability Status Scale (EDSS) from 1 to 6 (grade 6 includes patients with unilateral aid to ambulate)
* No contraindication for the administration of MP.
* Agree to participate in the study by means of a signed informed consent

Exclusion Criteria:

* Intake of anti-inflammatory steroids in the last 3 days.
* Patients with active bacterial, viral or fungal infections or undergoing treatment.
* Patients with hypertension.
* Patients with diabetes mellitus.
* Patients with hypo or hyperthyroidism.
* Patients with glaucoma.
* Patients with neoplasms.
* Diagnosis of systemic diseases such as: cardiovascular, pulmonary, hepatic, endocrine, gastrointestinal, etc.
* Patients with suspected or confirmed pregnancy by means of serum or urinary laboratory tests.
* Breastfeeding patients.
* Patients with a history of resistance to glucocorticoids.
* Patients with a history of severe adverse reactions to glucocorticoids.
* Patients with a history of hyposmia or anosmia.
* Patients diagnosed with active sinusitis.
* Patients with allergic rhinitis.
* Patients with upper respiratory tract infections.
* deviated septum
* History of nasal surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Patients' score on the Expanded Disability Status Scale (EDSS) before and after treatment to assess clinical efficacy of treatments | Days 0 and 30 after treatment
  * The Expanded Disability Status Scale has a minimum score of 0, when the patient has no MS-related disability or abnormalities, and a maximum score of 10, when death is caused by MS.
  * Patients will be assessed with the EDSS prior to treatment and 30 days after the treatment ends

SECONDARY OUTCOMES:
Concentration of inflammatory cytokines and chemokines in peripheral blood before, during, and after treatment | Days 0, 5 and 30 after treatment
  Enzyme-Linked Immunosorbent Assay (ELISA) to detect inflammatory molecules will be performed in plasma derived from blood samples taken from patients prior to treatment, on day 5 of treatment and 30 days after treatment

OTHER OUTCOMES:
Levels of lymphocyte subsets in peripheral blood before, during, and after treatment | Days 0, 5 and 30 after treatment
  •Flow cytometry will be performed using blood samples taken from patients prior to treatment, on day 5 of treatment and 30 days after treatment
Shannon and Chao1 indexes in feces samples to determine diversity and composition of intestinal microbiota in patients before and after treatment | Days 0 and 30 after treatment
  16S rRNA will be sequenced from isolated microbial DNA obtained from patient samples to determine global microbial composition prior to treatment and 30 days after treatment
Number of patients with adverse effects related to the methylprednisolone intranasal treatment as assessed by a questionnaire | Day 30 after treatment
  • The physician will assess possible adverse effects of the treatment using a questionnaire 30 days after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Neurología y Neurocirugía, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Information exchange for research purposes
Supporting Information: Study Protocol, CSR
Time Frame: Upon study completion, by request

DOCUMENTS (2):
  • Study Protocol (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT06223074/Prot_000.pdf
  • Informed Consent Form (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT06223074/ICF_001.pdf